CLINICAL TRIAL: NCT03228186
Title: Phase II Trial of Pevonedistat (TAK-924) Plus Docetaxel in Patients With Previously Treated Advanced Non-Small Cell Lung Cancer
Brief Title: Trial of Pevonedistat Plus Docetaxel in Patients With Previously Treated Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company discontinued the study drug.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.063; HUM00131436 (Other: University of Michigan)
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pevonedistat; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pevonedistat plus Docetaxel (Experimental): Pevonedistat 25mg/m2 days 1, 3, 5 Docetaxel 75mg/m2 day 1 21 day cycle
  Interventions: Drug: Pevonedistat; Drug: Docetaxel

INTERVENTIONS:
Drug: Pevonedistat — 25mg/m2 days 1, 3, 5
  Other Names: TAK-924
Drug: Docetaxel — 75mg/m2 day 1

SUMMARY:
This study is a single institution Phase II single arm trial to assess the efficacy of the combination of pevonedistat plus docetaxel in patients with previously treated advanced NSCLC (non-small cell lung cancer).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Histologically confirmed stage IV NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma, or not otherwise specified) or recurrent NSCLC not amenable to curative therapy
* Patients must have already received platinum-based chemotherapy; they may have also received prior immunotherapy or targeted therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.)
* Clinical laboratory values within appropriate parameters
* Female patients who are of childbearing potential and all males must agree to practice true abstinence or use effective methods of contraception
* Patients must be able to understand and sign the informed consent.
* Patients must have measurable disease as defined by RECIST v1.1 criteria
* It is preferable that patients have an adequate tissue sample available

Exclusion Criteria:

* Treatment with any investigational products within 4 weeks before the first dose of any study drug
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures
* Active uncontrolled infection or severe infectious disease, such as severe pneumonia, meningitis, or septicemia that require IV antibiotics within 2 weeks of starting study treatment
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period
* Diagnosed or treated for another malignancy within 2 years before randomization or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone resection.
* Life-threatening illness unrelated to cancer
* Patients with uncontrolled coagulopathy or bleeding disorder
* Known human immunodeficiency virus (HIV) seropositivity
* Known hepatitis B surface antigen seropositivity or known or suspected active hepatitis C infection
* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Known cardiopulmonary disease
* Uncontrolled high blood pressure (ie, systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)
* Prolonged rate corrected QT (QTc) interval ≥ 500 msec, calculated according to institutional guidelines
* Interstitial lung disease or pulmonary fibrosis
* Systemic antineoplastic therapy or radiotherapy for other malignant conditions within 14 days before the first dose of any study drug, except for hydroxyurea.
* Symptomatic or history of untreated brain or leptomeningeal metastases. Treated patients should be neurologically stable for 4 weeks after completion of appropriate therapy. Patients should be off steroids at least 3 days prior to start of therapy on clinical trial.
* Treatment with clinically significant metabolic enzyme inducers within 14 days before the first dose of the study drug. Clinically significant metabolic enzyme inducers are not permitted during this study (see Appendix III for more details).
* Female patients who are lactating, breastfeeding, or have a positive pregnancy test
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).
* Known hypersensitivity to docetaxel or other drugs formulated with polysorbate 80
* Prior therapy with docetaxel for non-small cell lung cancer
* Peripheral neuropathy of CTCAE v4.03 grade ≥ 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kalemkerian, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 patients screen failed
Period: Overall Study
Arm/Group | Pevonedistat Plus Docetaxel
Started | 31
Completed | 30
Not Completed | 1
Not completed — Patient never started treatment | 1

BASELINE CHARACTERISTICS:
Population: 9 patients were screen failed
Arm/Group | Pevonedistat Plus Docetaxel
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients That Respond to Treatment
Description: Response is defined as either Partial Response or Complete Response. Partial Response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.
  Complete Response is defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
Time Frame: Up to 2 Years
Population: 27 patients participated in the trial long enough to be considered evaluable for this outcome measure
Measure: Number (85% Confidence Interval); unit: percent of participants
Arm/Group | Pevonedistat Plus Docetaxel
Number analyzed (Participants) | 27
percent of participants | 22 [11 to 37]

2. Secondary Outcome: Median Progression Free Survival Time
Description: Progression-free survival is defined as the duration of time from start of treatment to time of progression.
  Progressive Disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Up to 2 Years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pevonedistat Plus Docetaxel
Number analyzed (Participants) | 27
days | 124 [88 to 209]

3. Secondary Outcome: Median Overall Survival Time
Description: Overall survival is defined as the duration of time from start of treatment to time of passing.
Time Frame: Up to 2 Years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pevonedistat Plus Docetaxel
Number analyzed (Participants) | 27
days | 397 [223 to NA] — The confidence interval for the median is calculated based on the confidence limits for the estimated survival function. If the upper limit does not cross the horizontal line at 0.5, then the upper confidence limit for the median does not exist.

4. Secondary Outcome: The Number of Patients Who Achieve Stable Disease
Description: Stable disease rate will be reported as the count and proportion of patients who achieve stable disease.
  Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for Partial Response (PR) nor sufficient increase to qualify for Progressive Disease (PD), taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Pevonedistat Plus Docetaxel
Number analyzed (Participants) | 27
Participants | 12

5. Secondary Outcome: The Number of Toxicities by System Organ Class
Description: All recorded toxicities will be listed and tabulated by system organ class. The NCI CTCAE version 4.03 will be utilized for AE reporting.
Time Frame: up to 30 days post last study drug dose, patients were allowed to stay on study drug treatment until progression. Data was collected over 3.5 years.
Population: Percentage of Grade 3-5 Adverse Events classified according to the Row Titles. The investigations group represents adverse events due to treatment drugs.
Measure: Number; unit: percentage of Grade 3-5 Adverse Events
Units Other Than Participants: adverse events
Arm/Group | Pevonedistat Plus Docetaxel
Number analyzed (Participants) | 30
Number analyzed (adverse events) | 90
percentage of Grade 3-5 Adverse Events
  Blood and Lymphatic system disorders- grade 3 | 10
  Gastrointestinal disorders- grade 3 | 6.7
  General disorders and administration site conditions- grade 3 | 10
  hepatobiliary disorders- grade 3 | 3.3
  infections and infestations- grade 3 | 3.3
  infections and infestations- grade 4 | 3.3
  investigations- grade 3 | 16.7
  investigations- grade 4 | 13.3
  metabolism and nutrition disorders- grade 3 | 3.3
  nervous system disorders- grade 3 | 3.3
  respiratory, thoracic and mediastinal disorders- grade 3 | 3.3
  Skin and subcutaneous tissue disorders- grade 3 | 3.3

ADVERSE EVENTS:
Time Frame: Up to 30 days post treatment for Serious Adverse Events and Other (Not Including Serious) Adverse Events. Data for serious and non serious adverse events was collected over 3.5 years., All-Cause Mortality was assessed for up to 3.5 years
Description: No patients died while within the Adverse Event Reporting windows
Arm/Group | Pevonedistat Plus Docetaxel
All-Cause Mortality (participants affected / at risk) | 24/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pevonedistat Plus Docetaxel (N=30)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis infection (Infections and infestations) | 1 (1)
fatigue (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hepatobiliary Disorders- other (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infections (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pevonedistat Plus Docetaxel (N=30)
Abdominal pain (General disorders) | 3 (4)
Alanine aminotransferase increased (Investigations) | 13 (24)
Alkaline phosphatase increased (Investigations) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Anemia (Investigations) | 5 (5)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 15 (23)
Back pain (General disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 2 (3)
Confusion (Psychiatric disorders) | 3 (4)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema limbs (General disorders) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 22 (28)
Fever (General disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematuria (Investigations) | 1 (1)
Hyperglycemia (Investigations) | 5 (5)
Hyperkalemia (Investigations) | 1 (1)
Hypertension (Cardiac disorders) | 2 (3)
Hypocalcemia (Investigations) | 1 (1)
Hypophosphatemia (Investigations) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 3 (5)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail infection (Infections and infestations) | 1 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (13)
Neutrophil count decreased (Investigations) | 7 (9)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 5 (5)
Pain in extremity (General disorders) | 5 (6)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (17)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Watering eyes (Eye disorders) | 4 (4)
Weight loss (Metabolism and nutrition disorders) | 4 (4)
White blood cell decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT03228186/Prot_SAP_ICF_000.pdf